CLINICAL TRIAL: NCT03670108
Title: Impact of Personalized SMS in Relay of Therapeutic Education Programs to Improve the Physical Activity of Patients in Rheumatology
Brief Title: "SMS - Heals My Health"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Cochin (Other)
Responsible Party: Principal Investigator, Serge Perrot, professor, Hôpital Cochin
Other Study IDs: 2016-A00580-51
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: to Help Improve the Quality of Life of Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients receiving an individualized SMS
- patients receiving a standard SMS

SUMMARY:
Therapeutic patient education is an approach that has shown its usefulness in rheumatology, but the duration of its impact is limited, and therapeutic revisions are regularly necessary. The practice of physical activity is one of the goals of TPE in rheumatology and new technologies, such as SMS messages represent a possible complementary tool to amplify behavioral changes The study primary objective is to evaluate the impact of individualized SMS compared to standard SMS messages on the physical activity of patients with chronic inflammatory rheumatism or osteoporosis, included in a therapeutic education program. Our hypothesis is that individualized SMS has a higher efficiency compared to standard SMS messages to increase the practice of physical activity in these patients.

ELIGIBILITY:
Inclusion Criteria:

* patient age from 18 to 75 years
* Participated in therapeutic patient education program osteoporosis disease and inflammatory rheumatism disease
* Having given their written consent
* French speaking
* Possessing a telephone tool that accepts SMS

Exclusion Criteria:

* Patients unable to read SMS for practical, linguistic or cognitive reasons
* Patients who can not, for medical reasons or disability, set up 30 minutes of moderate physical activity (walking or other moderate activity) per day
* Having already participated in a similar study in inflammatory rheumatism or osteoporosis
* Already having the required level of physical activity: performing more than 30 minutes of moderate physical activity (walking or other moderate activity)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with osteoporosis or inflammatory rheumatism aged between 18 and 75 years, who participated in the patient's therapeutic education program
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-02-12 (Estimated); Study Completion 2020-01-12 (Estimated)

PRIMARY OUTCOMES:
physical activity | 1 YEAR
  evaluate the percentage of patients reaching 30 minutes of moderate physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No